CLINICAL TRIAL: NCT04336488
Title: Effectiveness of Matrix Metalloproteinase Neutralizing Agent in Treatment of Oral Lichen Planus: A Pilot Study
Brief Title: Matrix Metalloproteinases Neutralizing Agents in Oral Lichen Planus
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jaylane kadry Ghonima (Other)
Responsible Party: Sponsor-Investigator, Jaylane kadry Ghonima, assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMPs in lichen
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Oral Lichen Planus
Keywords: matrix metalloproteinase inhibitors, orochem, OLP
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Matrix Metalloproteinase Inhibitors; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: double equal arms
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participant, investigator as well as outcome assessor are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Orochem (Test) (Experimental): fifteen patients with lichen planus will be treated with MMPs neutralizing agent 3 times daily for 3 weeks. then pain, discomfort and disease severity will be assessed at 1 and 3 weeks periods.
  Interventions: Drug: Matrix Metalloproteinase Inhibitors (Orochem)
- Conventional (Control) (Active Comparator): fifteen patients with oral lichen planus confirmed with a biopsy will be treated with topical corticosteroids, topical antifungal 3 timed daily for 3 weeks. then pain, discomfort and disease severity will be assessed at 1 and 3 weeks periods.
  Interventions: Drug: Kenacort A,

INTERVENTIONS:
Drug: Matrix Metalloproteinase Inhibitors (Orochem) — topical application of MMP inhibitors for 3 weeks to evaluate its effectiveness in treating oral lichen planus
  Arms: Orochem (Test)
Drug: Kenacort A, — topical application of both drugs 3 times daily for 3 weeks as an active control
  Other Names: miconaz gel
  Arms: Conventional (Control)

SUMMARY:
The current study will be conducted to evaluate the effectiveness of matrix metalloproteinases inhibitors on erosive oral lichen planus.

DETAILED DESCRIPTION:
Matrix metalloproteinases inhibitor (Orochem) will be given to patients with Oral erosive lichen planus three times daily for 3 weeks. Then the subjective discomfort and pain severity as well as the objective disease severity scores will be collected.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with erosive OLP confirmed with a biopsy.
* patients should have symptomatic lesions

Exclusion Criteria:

* Patients who were under anticoagulant medications, suffering from any systemic diseases or having any physical or mental abnormality, pregnant and lactating women, smokers.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
change in disease severity score | change in disease severity score from baseline to 3 weeks
  Thongprasom disease severity score (5-0)

CONTACTS AND LOCATIONS:
Overall Officials: Hossam H. AlSabbagh, As. lecturer, Principal Investigator — Alexandria University
Locations (1):
- periodontology department, Faculty of dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
participants data are not to be shared